CLINICAL TRIAL: NCT00411645
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Prophylactic Use of Maribavir for the Prevention of Cytomegalovirus Disease in Recipients of Allogeneic Stem Cell Transplants.
Brief Title: Prophylactic Use of Maribavir for the Prevention of Cytomegalovirus (CMV) Disease in Stem Cell Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1263-300; 2006-005692-18 (EudraCT Number); SHP620-300 (Other: Shire); NCT00430339 (obsolete NCT alias)
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Cytomegalovirus Infections
Keywords: prevention; prophylaxis; Cytomegalovirus; CMV; allogeneic stem cell transplant; SCT
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — maribavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: maribavir
- B (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: maribavir — 100 mg twice daily for up to 12 weeks
  Arms: A
Other: placebo — twice daily for up to 12 weeks
  Arms: B

SUMMARY:
The purpose of this research study is to investigate whether or not maribavir is safe and effective for preventing CMV disease when taken by mouth for up to 12 weeks in patients who have had a stem cell transplant.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) infections remain a significant problem following various types of transplants that are associated with strong immunosuppressive therapy. Maribavir is a new oral anti-CMV drug with a novel mechanism of action compared to currently available anti-CMV drugs. This study will test the safety and efficacy of maribavir for the prevention of CMV disease when given as prophylaxis for up to 12 weeks following allogeneic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic stem cell transplant recipient
* Recipient or donor CMV seropositive
* Have transplant engraftment
* Able to swallow tablets

Exclusion Criteria:

* CMV organ disease
* HIV infection
* Use of other anti-CMV therapy post-transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2006-12-13 (Actual); Primary Completion 2008-11-10 (Actual); Study Completion 2009-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (97):
- United States (56):
  - University of Arkansas Myeloma Institute, Little Rock, Arkansas
  - City of Hope Medical Center, Duarte, California
  - Scripps Green Hospital, La Jolla, California
  - UCSD Moores Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Shands Hospital, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - St Francis Hospital, Beech Grove, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University Medical Center University of Louisville Hospital, Louisville, Kentucky
  - Greenbaum Cancer Center, Baltimore, Maryland
  - Massachusettes General, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State Medical Center, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital,Weill Cornell Medical Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke Medical Center, Durham, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - The Jewish Hospital, Cincinnati, Ohio
  - Ireland Cancer Center Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Sciences University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson, Philadelphia, Pennsylvania
  - Jeanes Hospital - Temple, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Medical College of Virginia, Richmond, Virginia
  - VA Puget Sound Health Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
- Belgium (5):
  - ZNA Stuivenberg, Antwerp
  - AZ Sint Jan, Department of Hematology, Bruges
  - Cliniques Universitaires St,Luc Dept Hematology, Brussels
  - UZ Gasthuisberg, Leuven
  - CHU Sart -Tilman Department of Medicine, Hematology, Liège
- Canada (5):
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - McMaster University Medical Center, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa General Campus, Ottawa, Ontario
  - Hopital l'Enfant Jesus, Québec, Quebec
- France (6):
  - Hopital Henri Mondor, Créteil
  - Edouard Herriot Hopital, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Hotel Dieu, Nantes
  - Hopital St. Louis, Paris
  - Hopital Haut-Leveque, Pessac
- Germany (10):
  - Universitaetsklinikum Koeln, Clinic I for internal Medicine, Cologne
  - Univ. Clinic Dresden, Dresden
  - University Clinic of Dresden, Dresden
  - University of Essen, Essen
  - University of Freiburg, Freiburg im Breisgau
  - University of Hamburg-Eppendorf, Hamburg
  - Hannover, Medizinische Hochschule, Hanover
  - University of Heidelberg, Heidelberg
  - Johannes-Gutenberg University, Mainz
  - University Clinic of Ulm, Ulm
- Italy (5):
  - Careggi University Hospital, Florence
  - University of San Martino Hospital, Genova
  - San Raffaele del Monte Tabor, Milan
  - Pescara Hospital, Pescara
  - Bianchi-Melacrino-Morelli Hospital, Reggio Calabria
- Spain (3):
  - Barcelona Hospital, Barcelona
  - Duran i Reynals Hospital, Barcelona
  - University of Salamanca, Salamanca
- Sweden (4):
  - Karolinska University Hospital, Huddinge, Stockholm County
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital,Huddinge, Stockholm
  - Akademiska Sjukhuset, Dept Hematology, Uppsala
- United Kingdom (3):
  - University College Hospital, London
  - Royal Free Hospital, London
  - Hammersmith Hospital, London

REFERENCES:
- [Derived] Marty FM, Ljungman P, Papanicolaou GA, Winston DJ, Chemaly RF, Strasfeld L, Young JA, Rodriguez T, Maertens J, Schmitt M, Einsele H, Ferrant A, Lipton JH, Villano SA, Chen H, Boeckh M; Maribavir 1263-300 Clinical Study Group. Maribavir prophylaxis for prevention of cytomegalovirus disease in recipients of allogeneic stem-cell transplants: a phase 3, double-blind, placebo-controlled, randomised trial. Lancet Infect Dis. 2011 Apr;11(4):284-92. doi: 10.1016/S1473-3099(11)70024-X. Epub 2011 Mar 21. PMID 21414843

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo twice daily (BID) for up to 12 weeks.
- Maribavir 100 mg BID: Participants received maribavir 100 mg twice daily (BID) for up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Maribavir 100 mg BID
Started | 227 | 454
Completed | 146 | 290
Not Completed | 81 | 164
Not completed — Consent Withdrawn | 13 | 22
Not completed — Death | 56 | 135
Not completed — Investigator/Sponsor Decision | 10 | 7
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Maribavir 100 mg BID | Total
Number analyzed (Participants) | 227 | 454 | 681
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (13.1) | 49 (12.5) | 49 (12.7)
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 74 | 136 | 210
  45 to 64 years | 134 | 286 | 420
  65 to 75 years | 18 | 32 | 50
  > 75 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 189 | 287
  Male | 129 | 265 | 394

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Endpoint Committee (EC)-Confirmed Cytomegalovirus (CMV) Disease Within 6 Months Post-Transplantation
Description: All investigator-determined cases of CMV disease (i.e., CMV infection or CMV organ disease), were adjudicated by an independent, blinded EC. CMV infection was assessed by (1) pp65 antigenemia assay; (2) CMV DNA polymerase chain reaction (PCR); (3) either assay (pp65 antigenemia or CMV DNA PCR); or (4) initiation of anti-CMV therapy. CMV infection was defined as: CMV infection detected by a positive result from a CMV laboratory assay from at least one central laboratory assay (pp65 antigenemia or CMV DNA PCR assay in plasma) and fever >/=38 °C on >/=2 occasions >/=24 hours apart within a 7-day period and at least one of the following: new or increased malaise, two successive measurements of leucopenia (white blood cell [WBC] count <3500/mm3 or a WBC count decrease of 20% if the cell count prior to onset of clinical symptoms was >4000/mm3) >/=24 hours apart, atypical lymphocytosis >/=5%, and thrombocytopenia. CMV organ disease was defined as described by Ljungman et al., 2002.
Time Frame: 6 months post-transplant
Population: The Intent-to-Treat (ITT) population, defined as all participants who were randomized to one of the therapy groups, regardless of whether the participant received study drug or had any post-baseline evaluations.
Measure: Number; unit: participants
Arm/Group | Placebo | Maribavir 100 mg BID
Number analyzed (Participants) | 227 | 454
participants | 11 | 20
Statistical Analysis 1: Comparison: Placebo vs Maribavir 100 mg BID; Test type: Superiority or Other; p = 0.789, Cochran-Mantel-Haenszel — The p-value is from the Cochran-Mantel-Haenszel test, adjusting for recipient CMV serostatus (R+ or R-) and transplant type (myeloablative or non-myeloablative/reduced intensity); Odds Ratio (OR) = 0.902, 95% CI 2-sided [0.424 to 1.920] — Mantel-Haenszel odds ratio for maribavir versus placebo

2. Secondary Outcome: Number of Participants With CMV Infection or EC-confirmed CMV Disease Within 6 Months Post-transplant
Description: as for outcome 1
Time Frame: 6 months post-transplant
Population: The ITT population, defined as all participants who were randomized to one of the therapy groups, regardless of whether the participant received study drug or had any post-baseline evaluations.
Measure: Number; unit: participants
Arm/Group | Placebo | Maribavir 100 mg BID
Number analyzed (Participants) | 227 | 454
participants
  pp65 antigenemia assay | 88 | 143
  CMV DNA PCR assay | 77 | 152
  pp65 antigenemia or CMV DNA PCR assay | 101 | 183
  Initiation of anti-CMV therapy | 92 | 172
Statistical Analysis 1: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of pp65 antigenemia assay; Test type: Superiority or Other; p = 0.056, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.721, 95% CI 2-sided [0.515 to 1.008] — Mantel-Haenszel odds ratio for maribavir versus placebo
Statistical Analysis 2: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of CMV DNA PCR assay; Test type: Superiority or Other; p = 0.904, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.979, 95% CI 2-sided [0.697 to 1.375] — Mantel-Haenszel odds ratio for maribavir versus placebo
Statistical Analysis 3: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of pp65 antigenemia or CMV DNA PCR assay; Test type: Superiority or Other; p = 0.289, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.838, 95% CI 2-sided [0.606 to 1.161] — Mantel-Haenszel odds ratio for maribavir versus placebo
Statistical Analysis 4: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of initiation of anti-CMV therapy; Test type: Superiority or Other; p = 0.493, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.891, 95% CI 2-sided [0.640 to 1.239] — Mantel-Haenszel odds ratio for maribavir versus placebo

3. Secondary Outcome: Time to Onset of CMV Infection or EC-confirmed CMV Disease Within 6 Months Post- Transplantation
Description: All investigator-determined cases of CMV disease (i.e., CMV infection or CMV organ disease) were adjudicated by an independent, blinded EC. CMV infection was assessed by (1) pp65 antigenemia assay or (2) CMV DNA polymerase chain reaction (PCR). CMV infection was defined as: CMV infection detected by a positive result from a CMV laboratory assay from at least one central laboratory assay (pp65 antigenemia or CMV DNA PCR assay in plasma) and fever >/=38 °C on >/=2 occasions >/=24 hours apart within a 7-day period and at least one of the following: new or increased malaise, two successive measurements of leucopenia (white blood cell [WBC] count <3500/mm3 or a WBC count decrease of 20% if the cell count prior to onset of clinical symptoms was >4000/mm3) >/=24 hours apart, atypical lymphocytosis >/=5%, and thrombocytopenia. CMV organ disease was defined as described by Ljungman et al., 2002.
Time Frame: 6 months post-transplant
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Maribavir 100 mg BID
Number analyzed (Participants) | 227 | 454
days | 21 [5 to 22] | 22 [6 to 29]
Statistical Analysis 1: Comparison: Placebo vs Maribavir 100 mg BID; Test type: Superiority or Other; p = 0.129, Log Rank
Statistical Analysis 2: Comparison: Placebo vs Maribavir 100 mg BID; Test type: Superiority or Other; p = 0.130, Wald Chi-squared — The p-value from Wald Chi-Square test for treatment effect; Adjusted hazard ratio = 0.83, 95% CI 2-sided [0.65 to 1.06] — Maribavir versus placebo; based on Cox's proportional hazards regression model: time = recipient CMV serostatus (R+ or R-) + transplant type (myeloablative or non-myeloablative/reduced intensity) + treatment

4. Secondary Outcome: Number of Participants With Investigator-determined CMV Disease
Description: CMV infection was assessed by (1) pp65 antigenemia assay; (2) CMV DNA polymerase chain reaction (PCR); (3) either assay (pp65 antigenemia or CMV DNA PCR); or (4) initiation of anti-CMV therapy. CMV infection was defined as: CMV infection detected by a positive result from a CMV laboratory assay from at least one central laboratory assay (pp65 antigenemia or CMV DNA PCR assay in plasma) and fever >/=38 °C on >/=2 occasions >/=24 hours apart within a 7-day period and at least one of the following: new or increased malaise, two successive measurements of leucopenia (white blood cell [WBC] count <3500/mm3 or a WBC count decrease of 20% if the cell count prior to onset of clinical symptoms was >4000/mm3) >/=24 hours apart, atypical lymphocytosis >/=5%, and thrombocytopenia. CMV organ disease was defined as described by Ljungman et al., 2002.
Time Frame: Through 12 months post-transplant (Day 1 to 100 days, 6 months, and 12 months post-transplant)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Maribavir 100 mg BID
Number analyzed (Participants) | 227 | 454
participants
  100 days post-tranplant | 6 | 16
  6 months post-transplant | 11 | 26
  12 months post-transplant | 13 | 28
Statistical Analysis 1: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of 100 days post-transplant; Test type: Superiority or Other; p = 0.542, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of 6 months post-transplant; Test type: Superiority or Other; p = 0.637, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of 12 months post-transplant; Test type: Superiority or Other; p = 0.825, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With CMV Infection or EC-confirmed CMV Disease Within 100 Days Post-Transplantation
Description: as for outcome 1
Time Frame: 100 days post-transplant
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Maribavir 100 mg BID
Number analyzed (Participants) | 227 | 454
participants
  pp65 antigenemia assay | 79 | 120
  CMV DNA PCR assay | 69 | 126
  pp65 antigenemia assay or CMV DNA PCR assay | 92 | 157
  Initiation of anti-CMV therapy | 85 | 139
  EC-confirmed disease | 6 | 11
Statistical Analysis 1: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of pp65 antigenemia assay; Test type: Superiority or Other; p = 0.022, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.669, 95% CI 2-sided [0.474 to 0.946] — Mantel-Haenszel odds ratio for maribavir versus placebo
Statistical Analysis 2: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of CMV DNA PCR assay; Test type: Superiority or Other; p = 0.468, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.878, 95% CI 2-sided [0.617 to 1.247] — Mantel-Haenszel odds ratio for maribavir versus placebo
Statistical Analysis 3: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of pp65 antigenemia assay or CMV DNA PCR assay; Test type: Superiority or Other; p = 0.125, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.772, 95% CI 2-sided [0.555 to 1.075] — Mantel-Haenszel odds ratio for maribavir versus placebo
Statistical Analysis 4: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of initiation of anti-CMV therapy; Test type: Superiority or Other; p = 0.069, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.731, 95% CI 2-sided [0.521 to 1.026] — Mantel-Haenszel odds ratio for maribavir versus placebo
Statistical Analysis 5: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of EC-confirmed disease; Test type: Superiority or Other; p = 0.860, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.913, 95% CI 2-sided [0.332 to 2.508] — Mantel-Haenszel odds ratio for maribavir versus placebo

6. Secondary Outcome: Number of Participants With EC-confirmed CMV Disease Within 12 Months Post-Transplantation
Description: as for outcome 1
Time Frame: 12 months post-transplant
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Maribavir 100 mg BID
Number analyzed (Participants) | 227 | 454
participants | 13 | 22
Statistical Analysis 1: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of 12 months post-transplant; Test type: Superiority or Other; p = 0.617, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.835, 95% CI 2-sided [0.411 to 1.693] — Mantel-Haenszel odds ratio for maribavir versus placebo

7. Secondary Outcome: Percent of Participants With Acute Graft-Versus-Host Disease (GVHD)
Description: Analysis of acute GVHD was based on reported adverse events that mapped to the relevant MedDRA dictionary terms for acute GVHD. The percentage reported is for the occurrence of any grade of acute GVHD.
Time Frame: Through 6 months post-transplant (Days 1 to 100 and 6 months post-transplant)
Population: The ITT Safety (ITT-S) population, defined as participants in the ITT population who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Maribavir 100 mg BID
Number analyzed (Participants) | 223 | 451
percentage of participants
  100 days post-transplant | 39 | 40
  6 months post-transplant | 43 | 44
Statistical Analysis 1: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of 100 days post-transplant; Test type: Superiority or Other; p = 0.7808, Cochran-Mantel-Haenszel — The p-value is from the Cochran-Mantel-Haenszel test, adjusting for recipient CMV serostatus (R+ or R -) and transplant type (myeloablative or non-myeloablative/reduced intensity); Odds Ratio (OR) = 1.048, 95% CI 2-sided [0.754 to 1.457] — Mantel-Haenszel odds ratio for maribavir versus placebo
Statistical Analysis 2: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of 6 months post-transplant; Test type: Superiority or Other; p = 0.6946, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.068, 95% CI 2-sided [0.771 to 1.479] — Mantel-Haenszel odds ratio for maribavir versus placebo

8. Secondary Outcome: Percent of Participants With Chronic Graft-Versus-Host Disease (GVHD)
Description: Analysis of chronic GVHD was based on reported adverse events that mapped to the relevant MedDRA dictionary terms for chronic GVHD. The percentage reported is for the occurrence of any grade of chronic GVHD.
Time Frame: Through 6 months post-transplant (Days 1 to 100 and 6 months post-transplant)
Population: The ITT-S population, defined as participants in the ITT population who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Maribavir 100 mg BID
Number analyzed (Participants) | 223 | 451
percentage of participants
  100 days post-transplant | 5 | 6
  6 months post-transplant | 25 | 19
Statistical Analysis 1: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of 100 days post-transplant; Test type: Superiority or Other; p = 0.6304, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.186, 95% CI 2-sided [0.592 to 2.375] — Mantel-Haenszel odds ratio for maribavir versus placebo
Statistical Analysis 2: Comparison: Placebo vs Maribavir 100 mg BID; Analysis of 6 months post-transplant; Test type: Superiority or Other; p = 0.1019, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.726, 95% CI 2-sided [0.495 to 1.066] — Mantel-Haenszel odds ratio for maribavir versus placebo

9. Secondary Outcome: Number of Participants Who Died Within 12 Months Post-Transplantation
Time Frame: Through 12 months post-transplant (Days 1 to 100, 6 months, and 12 months post-transplant)
Population: The ITT-S population, defined as participants in the ITT population who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Maribavir 100 mg BID
Number analyzed (Participants) | 223 | 451
participants
  100 days post-transplant | 19 | 30
  6 months post-transplant | 37 | 88
  12 months post-transplant | 59 | 139

10. Secondary Outcome: Plasma Concentration of Maribavir During Treatment
Description: Pharmacokinetic (PK) profile sampling was performed to evaluate plasma concentrations of Maribavir. During the study drug administration period, blood samples for this purpose were collected on Day 7 (Week 1) and at Week 4. Every effort was made to ensure that doses were administered 12 hours apart on the day before and on the day of PK sampling. Permissible assessment windows for PK profile sampling purposes were +/- 3 days and +/- 5 days for the 1- and 4- week samples, respectively. Samples were analyzed by a validated liquid chromatography tandem mass spectrometry (LC/MS/MS) method. The validated lower limit of quantitation (LLOQ) in plasma was 0.2 μg/mL.
Time Frame: 12 hours post-dose after 1 and 4 weeks of treatment
Population: The pharmacokinetic (PK) population, defined as those participants in the ITT population from whom plasma samples were drawn, tested for maribavir concentrations, and complete, evaluable PK data were available.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Maribavir 100 mg BID
Number analyzed (Participants) | 66
μg/mL
  1 week post-dose, n=63 | 2.11 (2.10)
  4 weeks post-dose, n=48 | 2.19 (1.99)

11. Secondary Outcome: Plasma Concentration of Maribavir Metabolite VP 44469 During Treatment
Description: Pharmacokinetic (PK) profile sampling was performed to evaluate plasma concentrations of VP 44469, a metabolite of Maribavir. During the study drug administration period, blood samples for this purpose were collected on Day 7 (Week 1) and at Week 4. Every effort was made to ensure that doses were administered 12 hours apart on the day before and on the day of PK sampling. Permissible assessment windows for PK profile sampling purposes were +/- 3 days and +/- 5 days for the 1- and 4- week samples, respectively. Samples were analyzed by a validated liquid chromatography tandem mass spectrometry (LC/MS/MS) method. The validated lower limit of quantitation (LLOQ) in plasma was 0.2 μg/mL.
Time Frame: 12 hours post-dose after 1 and 4 weeks of treatment
Population: The PK population, defined as those participants in the ITT population from whom plasma samples were drawn, tested for maribavir concentrations, and complete, evaluable PK data were available.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Maribavir 100 mg BID
Number analyzed (Participants) | 66
μg/mL
  1 week post-dose, n=63 | 0.56 (0.36)
  4 weeks post-dose, n=48 | 0.65 (0.47)

ADVERSE EVENTS:
Description: Adverse events are reported for the ITT-S population, defined as participants in the ITT population who received at least one dose of study drug.
Arm/Group | Placebo | Maribavir 100 mg BID
Serious Adverse Events (participants affected / at risk) | 98/223 | 197/451
Other Adverse Events (participants affected / at risk) | 192/223 | 408/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=223) | Maribavir 100 mg BID (N=451)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Aplasia Pure Red Cell (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 | 4
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 0 | 1
Leukaemia Recurrent (Blood and lymphatic system disorders) | 6 | 15
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphoproliferative Disorder (Blood and lymphatic system disorders) | 1 | 5
Myelodysplastic Syndrome (Blood and lymphatic system disorders) | 2 | 1
Myeloma Recurrence (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Non-Hodgkin's Lymphoma Recurrent (Blood and lymphatic system disorders) | 4 | 5
Pancytopenia (Blood and lymphatic system disorders) | 1 | 4
Relapse of underlying disease (Blood and lymphatic system disorders) | 13 | 21 — Relapse of underlying disease includes the following MedDRA Preferred Terms: "Leukemia recurrent, myeloma recurrence, non-Hodgkin's lymphoma recurrent, and myelodysplastic syndrome"
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 0 | 2
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 2
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 3
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 3
Caecitis (Gastrointestinal disorders) | 0 | 2
Clostridium Difficile Colitis (Gastrointestinal disorders) | 3 | 5
Colitis (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Eosinophilic Colitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastroenteritis Caliciviral (Gastrointestinal disorders) | 0 | 1
Gastroenteritis Viral (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 2
Gingivitis (Gastrointestinal disorders) | 0 | 1
Helicobacter Gastritis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Lactose Intolerance (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4
Peritonitis Bacterial (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal Lesion (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5
Catheter Site Infection (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 2 | 2
Pyrexia (General disorders) | 14 | 28
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic Encephalopathy (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 3
Hepatitis Viral (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Venoocclusive Liver Disease (Hepatobiliary disorders) | 2 | 1
Acute Graft Versus Host Disease (Immune system disorders) | 25 | 56
Chronic Graft Versus Host Disease (Immune system disorders) | 1 | 1
Acinetobacter Bacteraemia (Infections and infestations) | 0 | 1
Adenovirus Infection (Infections and infestations) | 0 | 1
Aspergillosis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 3 | 9
Bacterial Sepsis (Infections and infestations) | 0 | 1
Bk Virus Infection (Infections and infestations) | 3 | 1
Catheter Sepsis (Infections and infestations) | 1 | 0
Central Line Infection (Infections and infestations) | 3 | 3
Cytomegalovirus Gastroenteritis (Infections and infestations) | 4 | 6
Cytomegalovirus Infection (Infections and infestations) | 4 | 10
Enterococcal Bacteraemia (Infections and infestations) | 1 | 1
Enterococcal Sepsis (Infections and infestations) | 0 | 2
Epstein-Barr Virus Infection (Infections and infestations) | 1 | 3
Escherichia Bacteraemia (Infections and infestations) | 1 | 0
Herpes Dermatitis (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Human Herpesvirus 6 Infection (Infections and infestations) | 1 | 0
Human Polyomavirus Infection (Infections and infestations) | 0 | 1
Klebsiella Bacteraemia (Infections and infestations) | 0 | 2
Klebsiella Sepsis (Infections and infestations) | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 1
Pneumonia Cytomegaloviral (Infections and infestations) | 1 | 6
Pseudomonal Bacteraemia (Infections and infestations) | 0 | 3
Salmonella Sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Serratia Bacteraemia (Infections and infestations) | 1 | 2
Staphylococcal Bacteraemia (Infections and infestations) | 3 | 9
Staphylococcal Sepsis (Infections and infestations) | 0 | 2
Streptococcal Bacteraemia (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Zygomycosis (Infections and infestations) | 1 | 2
Blood Stem Cell Transplant Failure (Injury, poisoning and procedural complications) | 1 | 3
Incision Site Infection (Injury, poisoning and procedural complications) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 1 | 3
Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 2
Blood Creatinine Increased (Investigations) | 1 | 1
Blood Uric Acid Increased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 3
International Normalised Ratio Increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure To Thrive (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Abscess (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy Steroid (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Compression Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Staphylococcal Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arachnoiditis (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 3
Extrapyramidal Disorder (Nervous system disorders) | 0 | 1
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 1
Meningitis Aseptic (Nervous system disorders) | 0 | 1
Meningitis Enterococcal (Nervous system disorders) | 1 | 0
Meningitis Viral (Nervous system disorders) | 0 | 1
Metabolic Encephalopathy (Nervous system disorders) | 1 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1
Subdural Haematoma (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 3
Dysuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 4 | 14
Renal Impairment (Renal and urinary disorders) | 0 | 2
Urinary Tract Infection (Renal and urinary disorders) | 2 | 2
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchopulmonary Aspergillosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Lung Infection Pseudomonal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Parainfluenzae Virus Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonia Fungal (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia Streptococcal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary Alveolar Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Syncytial Virus Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Catheter Thrombosis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 2
Microangiopathy (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 3
Syncope (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=223) | Maribavir 100 mg BID (N=451)
Anaemia (Blood and lymphatic system disorders) | 17 | 60
Neutropenia (Blood and lymphatic system disorders) | 18 | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 33
Abdominal Pain (Gastrointestinal disorders) | 17 | 34
Constipation (Gastrointestinal disorders) | 10 | 41
Diarrhoea (Gastrointestinal disorders) | 41 | 86
Dry Mouth (Gastrointestinal disorders) | 11 | 41
Dysgeusia (Gastrointestinal disorders) | 13 | 66
Dyspepsia (Gastrointestinal disorders) | 13 | 16
Nausea (Gastrointestinal disorders) | 33 | 68
Oral Candidiasis (Gastrointestinal disorders) | 10 | 34
Vomiting (Gastrointestinal disorders) | 27 | 48
Fatigue (General disorders) | 22 | 73
Oedema Peripheral (General disorders) | 28 | 58
Pyrexia (General disorders) | 28 | 46
Acute Graft Versus Host Disease (Immune system disorders) | 50 | 117
Bk Virus Infection (Infections and infestations) | 13 | 33
Staphylococcal Bacteraemia (Infections and infestations) | 15 | 17
Hepatic Enzyme Increased (Investigations) | 15 | 31
Weight Decreased (Investigations) | 29 | 41
Anorexia (Metabolism and nutrition disorders) | 11 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 30
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 26
Dizziness (Nervous system disorders) | 11 | 26
Headache (Nervous system disorders) | 21 | 44
Insomnia (Nervous system disorders) | 16 | 27
Tremor (Nervous system disorders) | 16 | 32
Renal Failure (Renal and urinary disorders) | 16 | 33
Urinary Tract Infection (Renal and urinary disorders) | 9 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 35
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 9 | 25
Erythema (Skin and subcutaneous tissue disorders) | 13 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 20
Rash (Skin and subcutaneous tissue disorders) | 30 | 59
Hypertension (Vascular disorders) | 13 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.